CLINICAL TRIAL: NCT05280548
Title: A Randomized, Open-label, Parallel-group, 18-month Phase 3 Study to Evaluate the Effect of Venglustat Compared With Usual Standard of Care on Left Ventricular Mass Index in Participants With Fabry Disease and Left Ventricular Hypertrophy
Brief Title: A Study to Evaluate the Effect of Venglustat Tablets on Left Ventricular Mass Index in Male and Female Adult Participants With Fabry Disease
Acronym: CARAT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC16158; U1111-1266-5068 (Registry Identifier: ICTRP); 2023-509715-91 (Registry Identifier: CTIS); 2021-002320-20 (EudraCT Number)
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — venglustat; agalsidase alfa; agalsidase beta; migalastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Venglustat (Experimental): Participants will receive venglustat once daily, orally
  Interventions: Drug: Venglustat (GZ402671)
- Standard of Care Therapy (Active Comparator): Participants will receive a locally approved Fabry therapy at the standard dose and schedule (in accordance with the locally approved prescribing information)
  Interventions: Drug: Agalsidase alfa; Drug: Agalsidase beta (GZ419828); Drug: Migalastat

INTERVENTIONS:
Drug: Venglustat (GZ402671) — Tablet; Oral
  Arms: Venglustat
Drug: Agalsidase alfa — Concentrate for solution for infusion; IV infusion
  Other Names: Replagal®
  Arms: Standard of Care Therapy
Drug: Agalsidase beta (GZ419828) — Powder for concentrate for solution for infusion; IV infusion
  Other Names: Fabrazyme®
  Arms: Standard of Care Therapy
Drug: Migalastat — Hard capsules; Oral
  Other Names: Galafold®
  Arms: Standard of Care Therapy

SUMMARY:
This is an 18-month, multicenter, randomized, active-control, parallel-group Phase 3 study, in which participants will be randomized to venglustat versus standard of care therapy (agalsidase alfa, agalsidase beta, or migalastat) to evaluate the effect of venglustat on left ventricular mass index (LVMI) in adult participants with Fabry disease and left ventricular hypertrophy.

* Study visits will take place approximately every 3 to 6 months
* Participants who complete the randomized period may continue to the long-term extension (LTE) to receive venglustat for up to additional 45 months with the total study duration up to 5.3 years maximum.

DETAILED DESCRIPTION:
Randomized period: the total duration will be up to approximately of 20 months (1 month screening 18 months of treatment and a possible follow-up period of 1 month if no participation in the long-term extension period)

Long-term extension period: the total duration will be from minimum 19 months (18 months of treatment and 1 month of follow-up period) to maximum 46 months (45 months of treatment and 1 month of follow-up period). The maximum total study duration is approximately 5.3 years

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 to 65 with previously confirmed diagnosis of Fabry disease and a history of clinical symptoms of Fabry disease.
* Participants may be receiving treatment with agalsidase alfa, agalsidase beta, or migalastat, or may be untreated.
* Left ventricular hypertrophy.
* Contraception for male or female participants: not pregnant or breastfeeding; no sperm donating for male participant.
* A signed informed consent must be provided prior to any study-related procedures.

Exclusion Criteria:

* History of transient ischemic attack, stroke, myocardial infarction, heart failure, major cardiovascular surgery or kidney transplantation.
* History of seizures currently requiring treatment.
* Underlying medical condition that may cause or contribute to left ventricular hypertrophy.
* Asymmetric hypertrophy by cardiac MRI at screening if considered by central reader to be not related to Fabry disease.
* Advanced cardiac fibrosis, defined as significant late gadolinium enhancement affecting 3 or more segments involving >50% of myocardial thickness on screening cardiac MRI.
* History of clinically significant cardiac arrhythmia. Atrial fibrillation that is well controlled on a stable medical regimen for at least 12 months is not an exclusion if the CHA2DS2-VASc score is 0 for males or 1 for females.
* Estimated glomerular filtration rate <45 mL/min/1.73m2.
* Presence of severe depression as measured by Beck's Depression Inventory (BDI)-II >28 and/or a history of an untreated, unstable major affective disorder within 1 year of the screening visit.
* Patients with hepatitis C, HIV, or hepatitis B infection.
* Positive SARS-CoV-2 virus test within 2 weeks of enrollment, or COVID-19 requiring hospitalization within 6 months of enrollment.
* History of drug and/or alcohol abuse.
* Moderate to severe hepatic impairment.
* History of or active hepatobiliary disease.
* Liver enzymes (alanine aminotransferase/aspartate aminotransferase) or total bilirubin >2 times the upper limit of normal.
* Strong or moderate inducers or inhibitors of cytochrome P450 CYP3A4 within 14 days or 5 half-lives, whichever is longer, prior to randomization.
* Known contraindication to undergoing MRI or known hypersensitivity to gadolinium-based contrast agents.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-12-06 (Estimated)

PRIMARY OUTCOMES:
Slope of left ventricular mass index as measured by cardiac magnetic resonance imaging (MRI) (central reading) | from baseline to 18 months

SECONDARY OUTCOMES:
Slope of estimated glomerular filtration rate (eGFR) as assessed by the chronic kidney disease epidemiology collaboration (CKD-EPI) creatinine equation | from baseline to 18 months
Change in T1 relaxation time, measured by cardiac MRI (central reading) | from baseline to 18 months
Change in global longitudinal strain, measured by echocardiography (central reading) | from baseline to 18 months
Percent Change in tiredness component of FD-PRO | from baseline to 18 months
Percent Change in swelling in lower extremities component of FD-PRO | from baseline to 18 months
Number of participants with adverse event (AE) and serious adverse event (SAE) | from baseline to 18 months
Change in Beck Depression Inventory-II (BDI-II) score | from baseline to 18 months
Change in the lens clarity by ophthalmological examination | from baseline to 18 months
Plasma venglustat concentrations at prespecified visits over the study duration | from baseline to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations Clinical Sciences and Operations, Study Director — Sanofi
Locations (54):
- United States (8):
  - University of Alabama -The Kirklin Clinic- Site Number : 8400010, Birmingham, Alabama
  - University of California Los Angeles Medical Center- Site Number : 8400008, Los Angeles, California
  - Emory University School of Medicine - Atlanta- Site Number : 8400009, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago- Site Number : 8400005, Chicago, Illinois
  - Maryam Banikazemi, MD- Site Number : 8400001, Hawthorne, New York
  - Renal Disease Research Institute- Site Number : 8400012, Dallas, Texas
  - University of Utah Health Hospital- Site Number : 8400006, Salt Lake City, Utah
  - Lysosomal and Rare Disorders Research and Treatment Center (LDRTC)- Site Number : 8400004, Fairfax, Virginia
- Investigational Site Number : 0400001, Graz, Austria
- Canada (4):
  - Investigational Site Number : 1240003, Calgary, Alberta
  - Investigational Site Number : 1240006, Edmonton, Alberta
  - Investigational Site Number : 1240002, Vancouver, British Columbia
  - Investigational Site Number : 1240005, Toronto, Ontario
- China (5):
  - Investigational Site Number : 1560002, Beijing
  - Investigational Site Number : 1560005, Beijing
  - Investigational Site Number : 1560001, Chengdu
  - Investigational Site Number : 1560007, Guangzhou
  - Investigational Site Number : 1560003, Shanghai
- Investigational Site Number : 2030001, Prague, Czechia
- Investigational Site Number : 2080001, Copenhagen, Denmark
- Investigational Site Number : 2500001, Garches, France
- Germany (4):
  - Investigational Site Number : 2760003, Berlin
  - Investigational Site Number : 2760004, Hochheim am Main
  - Investigational Site Number : 2760005, Mainz
  - Investigational Site Number : 2760001, Würzburg
- Greece (3):
  - Investigational Site Number : 3000002, Athens
  - Investigational Site Number : 3000003, Athens
  - Investigational Site Number : 3000001, Heraklion
- Italy (4):
  - Investigational Site Number : 3800001, Milan, Lombardy
  - Investigational Site Number : 3800002, Naples, Napoli
  - Investigational Site Number : 3800003, Naples, Napoli
  - Investigational Site Number : 3800004, Bologna
- Japan (7):
  - Investigational Site Number : 3920006, Sapporo, Hokkaido
  - Investigational Site Number : 3920007, Kagoshima, Kagoshima-ken
  - Investigational Site Number : 3920003, Kagoshima, Kagoshima-ken
  - Investigational Site Number : 3920005, Kawasaki, Kanagawa
  - Investigational Site Number : 3920002, Sendai, Miyagi
  - Investigational Site Number : 3920004, Fukuoka
  - Investigational Site Number : 3920001, Tokyo
- Investigational Site Number : 5280001, Amsterdam, Netherlands
- Investigational Site Number : 5780001, Bergen, Norway
- Poland (2):
  - Investigational Site Number : 6160003, Lodz, Lódzkie
  - Investigational Site Number : 6160001, Krakow
- South Korea (2):
  - Investigational Site Number : 4100002, Yangsan, Gyeongsangnam-do
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
- Spain (3):
  - Investigational Site Number : 7240002, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240003, Alicante
  - Investigational Site Number : 7240001, Pontevedra
- Taiwan (2):
  - Investigational Site Number : 1580003, Taichung
  - Investigational Site Number : 1580001, Taipei
- Turkey (Türkiye) (3):
  - Investigational Site Number : 7920001, Ankara
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920003, İzmit
- Investigational Site Number : 8260001, London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org